CLINICAL TRIAL: NCT03516591
Title: A Phase 1, Multicenter, Open Label Study of AMV564, a Bispecific CD33/CD3 T-cell Engager, in Patients With Intermediate or High-Risk Myelodysplastic Syndromes
Brief Title: A Phase 1 Study of AMV564 in Patients With Intermediate or High-Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amphivena Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AMV564-201
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Electron Transport Complex IV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (3+3 design) (Experimental): A 3 + 3 design, with dose-escalation of AMV564, up to a Maximum Tolerated Dose (MTD) level. AMV564 will be tested as a 14-Day CIV regimen (14-Day Continuous Intravenous Infusion Regimen).
  Interventions: Drug: AMV564 14-Day CIV
- Dose Expansion (Experimental): Following determination of the MTD of AMV564, the study will expand at the MTD or a dose level lower than the MTD to obtain initial estimates of response rates and additional information on safety.
  Interventions: Drug: AMV564 14-Day CIV

INTERVENTIONS:
Drug: AMV564 14-Day CIV — A 14-Day Continuous Intravenous Infusion regimen

SUMMARY:
An open label, Phase 1, study of AMV564 as monotherapy to assess the safety and efficacy in patients with Myelodysplastic Syndromes

DETAILED DESCRIPTION:
A dose-escalation with expansion study of AMV564 (T cell engager) as monotherapy in patients with intermediate-2 or high-risk Myelodysplastic Syndromes

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosis of MDS according to WHO 2016 criteria
* ECOG performance status of 0 or 1
* Intermediate-2 or high-risk disease per IPSS
* Fewer than 20% blasts in the bone marrow or peripheral blood
* Disease that is refractory to or relapsed from either a hypomethylating agent (e.g. decitabine or azacitidine) or a standard AML-type intensive regimen
* Adequate organ function
* Prior allogeneic transplant performed ≥ 3 months prior to first dose of AMV564 is allowed provided there is no evidence of active graft-versus-host disease (GVHD) and the patient has been off immunosuppressive therapy for ≥ 4 weeks.

Exclusion Criteria:

* History of, or known, central nervous system (CNS) disease involvement, or prior history of National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) Grade ≥ 3 drug-related CNS toxicity
* Prior allogeneic transplant if performed < 3 months prior to first dose of AMV564, if patient has active GVHD, or if patient has not been off immunosuppressive
* Prior treatment with a therapeutic agent targeting CD33 (e.g. gemtuzumab ozogamicin, SGN-CD33A or AMG 330).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (Dose Escalation) | DLTs will be evaluated through 28 days for the 14-Day Continuous Intravenous Infusion Infusion regimen, and 35 days for the Intermittent Intravenous Dosing regimen
  Dose limiting toxicity to be measured by AEs and SAEs by dose level
Overall Response Rate (Dose Expansion) | The treatment period will extend from initiation of AMV564 treatment until the Safety Follow Up visit (30 days after the end of infusion), or response assessment of the last induction cycle, whichever occurs later.
  Overall response rate (ORR), defined as the proportion of patients who achieve a CR, marrow CR or PR by IWG criteria. Point estimates for ORR, along with the approximate lower 1-sided 90% confidence intervals, will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Chun, MD, Study Director — Amphivena Therapeutics, Inc.
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - Washington University, Siteman Cancer Center, St Louis, Missouri
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided